CLINICAL TRIAL: NCT06126666
Title: A Phase 1 Dose Escalation and Expansion Study of ABL103, a Bispecific Antibody of 4-1BB and B7-H4, as a Single Agent in Subjects With Any Progressive Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study With ABL103 in Subjects With Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ABL Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABL103-1001
Record Dates: First submitted 2023-11-02; First posted 2023-11-13 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABL103 (Experimental): ABL103 will be administered biweekly of every 28-day cycle in the dose-escalation. The dosing interval to be used in tumor-expansion part will be evaluated based on the emerging safety and PK data from the dose-escalation part of the study.
  Interventions: Drug: ABL103

INTERVENTIONS:
Drug: ABL103 — ABL103 will be administered biweekly of every 28-day cycle in the dose-escalation. The dosing interval to be used in tumor-expansion part will be evaluated based on the emerging safety and PK data from the dose-escalation part of the study.

SUMMARY:
This is a first-in-human Phase 1, single-arm, open-label, multicenter, multiple-dose, dose-escalation study of ABL103 to evaluate the safety, tolerability, MTD (maximum tolerated dose) and/or RP2D (recommended phase 2 dose), pharmacokinetics, immunogenicity, preliminary antitumor activity of ABL103 in subjects with any progressive locally advanced(unresectable) or metastatic solid tumor who are relapsed or refractory following the last line of treatment and have no available standard of care option. This study includes 2 parts: a dose-escalation part and tumor-expansion part

ELIGIBILITY:
Inclusion Criteria:

* Subject must understand and be willing to provide informed consent and be able to comply with the study procedures and restrictions.
* Subject must be ≥18 years of age on the day of signing the informed consent form (ICF)
* Subject must have a histologically confirmed locally advanced unresectable, or metastatic solid tumor.
* Subject must be relapsed or be refractory to available standard therapy or they must be intolerant of available standard therapy.
* Subject must meet Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Subject must have an estimated life expectancy of at least 12 weeks.
* Subjects must be recovered from AEs from prior therapy to Grade 1 or the baseline grade more than 14 days prior to the first administration of the study drug, except alopecia or Grade 2 toxicities that are deemed stable or irreversible (eg, peripheral neuropathy)
* Subjects must have adequate hematologic, renal, hepatic, and thyroid functions confirmed based on the screening laboratory test within 7 days prior to the first administration of ABL103.

Exclusion Criteria:

* Subject has received prior anticancer monoclonal antibody treatment or investigational therapy within 28 days prior to the first administration of study drug.
* Subject has received prior chemotherapy or radiation therapy within 2 weeks or targeted small molecule therapy within 5 half-lives prior to the first administration of study drug.
* Subject requires or has received systemic steroid therapy or any other immunosuppressive therapy within 14 days prior to study drug administration.
* Subject has a history of drug-induced pneumonitis (interstitial lung disease) or currently has pneumonitis.
* Subject has risk factors for bowel obstruction or bowel perforation, including, but not limited to a history of acute diverticulitis, intra-abdominal abscess, and abdominal carcinomatosis.
* Subject discontinued from prior immunomodulatory therapy due to any intolerable immune-related adverse events (irAEs) requiring systemic steroid treatment.
* Subject has received prior treatment with anti-B7-H4 antibody and/or anti-4-1BB antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with Dose-Limiting Toxicities (DLT) | From Day 1 until disease progression or Day 28
  Number of subjects with Dose-Limiting Toxicities (DLT)
Number of subjects with Treatment-emergent Adverse Events (AEs), Serious Adverse Events (SAEs) and immune-related Adverse Events (irAEs) | From Day 1 until confirmed Complete Response (CR), disease progression, initiation of a new anticancer therapy, unacceptable toxicity, or subject's consent withdrawal, or investigator's decision to discontinue treatment, which came first
  Number of subjects with Treatment-emergent AEs, SAEs and irAEs
Number of subjects with Treatment-emergent Infusion related reactions (IRRs) | From Day 1 until confirmed CR, disease progression, initiation of a new anticancer therapy, unacceptable toxicity, or subject's consent withdrawal, or investigator's decision to discontinue treatment, which came first
  Number of subjects with Treatment-emergent IRRs
Number of subjects with the changes from baseline in laboratory values | From Day 1 until confirmed CR, disease progression, initiation of a new anticancer therapy, unacceptable toxicity, or subject's consent withdrawal, or investigator's decision to discontinue treatment, which came first
  Number of subjects with the changes from baseline in laboratory values

SECONDARY OUTCOMES:
Pharmacokinetic profile of ABL103 | From Day 1 until confirmed CR, disease progression, initiation of a new anticancer therapy, unacceptable toxicity, or subject's consent withdrawal, or investigator's decision to discontinue treatment, which came first, assessed up to 24 months
  serum concentration of ABL103 will be collected and analyzed to evaluate the PK of ABL103

CONTACTS AND LOCATIONS:
Overall Officials: Sangmi Lee, Study Director — Clinical development team
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam, Seoul
  - Seoul National University Hospital, Seoul, Seoul
  - Sevrance Hospital, Seoul, South Korea